CLINICAL TRIAL: NCT03275519
Title: Randomized Trial of Antibiotic Prophylaxis for Prevention of Symptomatic UTI in Stented, Distal Hypospadias Repair
Brief Title: Antibiotic Use in Distal Hypospadias Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 203532
Record Dates: First submitted 2017-08-11; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Hypospadias
Keywords: distal hypospadias repair; urinary tract infection; prophylactic antibiotic use
MeSH Terms: conditions — Hypospadias; Urinary Tract Infections

STUDY DESIGN:
Intervention Model Description: Using the block randomization procedures, a subject was assigned to a study group by computer using the REDCap randomization module. Subjects were randomized to receive post operative antibiotics or to not receive any antibiotics postoperative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics prophylaxis cohort (Active Comparator): Subjects were prescribed prophylactic antibiotics after the hypospadias surgery.
  Interventions: Other: Randomization to receive prophylactic antibiotics after surgery
- Antibiotic-sparing cohort (Active Comparator): Subjects were not prescribed prophylactic antibiotics after the hypospadias surgery.
  Interventions: Other: Randomization to not receive prophylactic antibiotics after surgery.

INTERVENTIONS:
Other: Randomization to not receive prophylactic antibiotics after surgery. — No antibiotics were ordered after surgery.
  Arms: Antibiotic-sparing cohort
Other: Randomization to receive prophylactic antibiotics after surgery — In general, the antibiotic given is a combination sulfamethoxazole/ trimethoprim oral suspension (2-3 mg trimethoprim/kg by mouth once a day); or if indicated, nitrofurantoin (1mg/kg by mouth once daily). All subjects did not receive intraoperative antibiotics.
  Arms: Antibiotics prophylaxis cohort

SUMMARY:
Hypospadias is a common condition where the opening of the penis is not located at the tip, but along the underside of the penis. It is estimated to occur in 1/300 live male births, making it one of the most common birth defects. Degrees of hypospadias ranged from minor to severe depending on the location of the opening. Surgical repair is often required and involves placement of a catheter for the urine to drain with known urinary colonization found on prior retrospective studies. The current practice of using preventative antibiotics as long as the catheter is in place is conflicting with resent studies that show antibiotics may not be necessary to prevent urinary tract infections (UTIs).

The purpose of this study was to see how common symptomatic UTIs were after hypospadias repair surgery; and to see whether routine antibiotic use after surgery affected the rate of UTIs. Subjects were randomized to either receive antibiotics or no antibiotics after distal hypospadias repair. The research coordinator made follow-up phone calls with the family and the primary care provider (PCP) after stent removal, 30 days post surgery and after the 3 month post surgical visit.

DETAILED DESCRIPTION:
Males undergoing distal hypospadias repair involving stent placement were randomized to either receive or not to receive antibiotics post-operative. All subjects did not receive intra-operative antibiotics. Routine follow-up included having the stent removed one week post-op and a return visit at 3 months. The research nurse made follow-up phone calls to the family or the (PCP) one week after the stent was removed and at one month post-op to see how things were going with the child and again after teh 3 month post surgical visit, if the subject did not return after multiple rescheduling attempts.

ELIGIBILITY:
Inclusion Criteria:

* Males undergoing primary distal hypospadias repair with open urethral stent drainage.

Exclusion Criteria:

* Males undergoing fistula repair or glandular hypospadias repair without incontinent urethral stent drainage and hypospadias repair of mid or more proximal degrees of hypospadias were excluded from this study.

Ages: 3 Months to 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Males undergoing hypospadias repair on their penis.
Enrollment: 48 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of symptomatic UTI within 30 days post-surgery | 30 days post surgery
  Assess the prevalence of symptomatic UTI in subjects receiving standard of care dispensation of prophylaxis versus subjects selected to an antibiotic-sparing cohort.

SECONDARY OUTCOMES:
Evaluation of surgical site infections (SSIs) and complications of hypospadias repair | Approximately post surgery: 2 weeks (stent is in approximately 1 week and then 1 week after the stent is removed); 30 days; and 3 months
  Surgical site infections (SSIs) are measured using physical assessments at the stent removal visit. Complications of hypospadias repair (urethral fistula, meatal stenosis, dehiscence, and diverticulum) are measured using physical assessments at the stent removal visit and/or contact with the family or the PCP office 1 week after the stent removal; at the 30 day post operative time point; and at the 3 month follow-op visit.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Canon, Principal Investigator — Arkansas Children's Hospital, Pediatric Urology
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No